CLINICAL TRIAL: NCT04499274
Title: The Effect of an Ondansetron on Blood Coagulation: In Vitro, Volunteer Study Using Rotational Thromboelastometry
Brief Title: Ondansetron and Blood Coagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B-2008/631-305
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 ng/ml (Experimental): Blood specimen which was added 0 ul of ondansetron
  Interventions: Drug: 0 ul of ondansetron
- 200 ng/ml (Experimental): Blood specimen which was added 0.20 ul of ondansetron
  Interventions: Drug: 0.2 ul of ondansetron
- 2000 ng/ml (Experimental): Blood specimen which was added 2 ul of ondansetron
  Interventions: Drug: 2 ul of ondansetron
- 20000 ng/ml (Experimental): Blood specimen which was added 20 ul of ondansetron
  Interventions: Drug: 20 ul of ondansetron

INTERVENTIONS:
Drug: 0 ul of ondansetron — Venous blood is taken from 12 healthy volunteers and divided into four specimen bottles, which were added with different doses (0 nl) using ondansetron
  Arms: 0 ng/ml
Drug: 0.2 ul of ondansetron — Venous blood is taken from 12 healthy volunteers and divided into four specimen bottles, which were added with different doses (0.2 ul) using ondansetron
  Arms: 200 ng/ml
Drug: 2 ul of ondansetron — Venous blood is taken from 12 healthy volunteers and divided into four specimen bottles, which were added with different doses (2 ul) using ondansetron
  Arms: 2000 ng/ml
Drug: 20 ul of ondansetron — Venous blood is taken from 12 healthy volunteers and divided into four specimen bottles, which were added with different doses (20 ul) using ondansetron
  Arms: 20000 ng/ml

SUMMARY:
Ondansetron may alter whole blood coagulation. However, little is known about the dose-response relationships according to the blood concentration of ondansetron. The investigators therefore will perform the present study to measure the effect of ondansestron on the blood coagulation pathway according to the drug concentration level using a thromboelastography test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy vonlunteers
* Age: 20 to 65 years
* Body weight > 50 kg
* Volunteers who provided informed consent

Exclusion Criteria:

* Hematologic disease
* Anticoagulant medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Citrated Functional Fibrinogen | During the thromboelastography analysis/ an average of 1 hour
  Provides clot strength based on fibrinogen contribution

SECONDARY OUTCOMES:
Citrated Kaolin | During the thromboelastography analysis/ an average of 1 hour
  Normal thromboelastography
Citrated Kaolin Heparinase | During the thromboelastography analysis/ an average of 1 hour
  To assess the effect of heparin
Citrated Rapid Thromboelastography | During the thromboelastography analysis/ an average of 1 hour
  A quicker assessment of clot strength, without assessment of clot initiation
Heparinized Kaolin Heparinase | During the thromboelastography analysis/ an average of 1 hour
  To measure the platelet function
Activator F | During the thromboelastography analysis/ an average of 1 hour
  To eliminate the platelet function
Adenosine diphosphate | During the thromboelastography analysis/ an average of 1 hour
  To masure the drug effect
Arachidonic acid | During the thromboelastography analysis/ an average of 1 hour
  To masure the drug effect

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea